CLINICAL TRIAL: NCT01549743
Title: Clinical Trial to Assess the Pharmacokinetic Interaction Between Celecoxib and Rebamipide in Healthy Male Volunteers
Brief Title: The Pharmacokinetic Interaction Between Celecoxib and Rebamipide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HL-CER-101
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Celecoxib; rebamipide

ARMS (3):
- Celecoxib (Experimental)
  Interventions: Drug: Celecoxib
- Rebamipide (Experimental)
  Interventions: Drug: Rebamipide
- Celecoxib plus Rebamipide (Experimental)
  Interventions: Drug: Celecoxib plus Rebamipide

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 200mg will be administered orally twice a day for 3 days
  Arms: Celecoxib
Drug: Rebamipide — Rebamipide 100mg will be administered orally three times a day for 3 days
  Arms: Rebamipide
Drug: Celecoxib plus Rebamipide — Celecoxib plus Rebamipide same way as "arm: celecoxib" and "arm: rebamipide"
  Arms: Celecoxib plus Rebamipide

SUMMARY:
This clinical trial aims to assess the pharmacokinetic interaction between celecoxib and rebamipide in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ae least 50kg and BMI(body mass index) within the range of 18 to 27kg/m2
* Agreement with written informed consent

Exclusion Criteria:

* Subject with symptoms of acute disease within 28days prior to study medication dosing
* Subject with known for history which affect on the absorption, distribution, metabolism, excretion of drug
* Subject with clinically significant active cardiovascular, respiratory, renal, endocrine, hematologic, gastrointestinal, neurologic, autoimmunologic disease or malignant tumor
* Subject with unsuitable clinical test through the medical checkup(medical history, physical examination, ECG, laboratory test) within 28days prior to study medication dosing
* Subject with any of the following findings; i. AST(sGOT) or ALT(sGPT) > 1.5 fold normal value or ii. Total bilirubin > 1.5 fold normal value
* Subject with clinically significant allergic disease (except for mild allergic rhinitis, mild allergic dermatitis seems to be not need for medication)
* Subject with known for hypersensitivity reaction to celecoxib, rebamipide, sulphonamide analog
* Subject with asthma, acute rhinitis, nasal polyp, angioedema, urticaria, allergic reaction to aspirin or any other NSAIDs(including COX-2 inhibitors)
* Subject with hereditary disorders such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Use of any prescription medication within 14 days prior to study medication dosing
* Use of any medication(Over-the-counter medication, oriental medication, vitamin) within 7 days prior to study medication dosing
* Subject who has been taken meal which affect on the absorption, distribution, metabolism, excretion of drug
* Subject who is not able to taking the institutional standard meal
* Whole blood donation within 60days, component blood donation within 20days or receiving blood transfusion within 30days prior to study medication dosing
* Participation in any clinical investigation within 60days prior to study medication dosing
* Continued excessive use of caffeine (caffeine > five cups/day), alcohol(alcohol>30g/day) and severe heavy smoker(cigarette > 10 cigarettes per day)
* An impossible one who participate in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2012-06-13 (Actual); Study Completion 2012-06-13 (Actual)

PRIMARY OUTCOMES:
Cmax,ss, Cmin,ss, Tmax,ss, Cav,ss, AUCτ, DOF(= (Cmax-Cmin)/Cav), Swing | Day1(0hr), Day2 (0hr), Day3 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48hr)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, Ph.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- The Korea Univertisy Anam Hospital, Seoul, South Korea